CLINICAL TRIAL: NCT02687425
Title: Phase 2 Study to Assess the Safety and Efficiency of Pioglitazone in Combination With Imatinib Mesylate to Treat Chronic Phase Chronic Myelogenous Leukemia Patients
Brief Title: Safety and Efficiency Study of Pioglitazone in Combination With Imatinib Mesylate to Treat Chronic Myelogenous Leukemia
Acronym: SESPI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meng Li (Other)
Responsible Party: Sponsor-Investigator, Meng Li, professor, department of hematology, Wuhan Tongji Hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML-201602
Record Dates: First submitted 2016-01-27; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: Pioglitazone; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Pioglitazone; Imatinib Mesylate; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pioglitazone (Experimental): The patients under the long-term treatment of imatinib mesylate acquire pioglitazone additionally.
  Interventions: Drug: Pioglitazone; Drug: imatinib mesylate

INTERVENTIONS:
Drug: Pioglitazone — 15mg/day,po
  Other Names: Actos
Drug: imatinib mesylate — 400mg/day,po
  Other Names: tyrosine kinase inhibitors

SUMMARY:
The purpose of this study is to assess the safety and efficiency of adding pioglitazone to chronic phase chronic myelogenous leukemia patients having received imatinib mesylate who have acquired a stable molecular response but not complete molecular response.

DETAILED DESCRIPTION:
Although tyrosine-kinase inhibitors have profoundly converted the outcomes of chronic myelogenous leukemia patients ,the most of who could have a complete cytogenetic response, a large majority of patients could not come to a complete molecular response that is undetectable in breakpoint cluster region-Abelson chimeric oncogene transcripts. According to some previous researches, pioglitazone may target leukemia stem cells and induce them into cell cycle making them exit from quiescent undivided states. Subsequently, pioglitazone may gradually erode leukemia stem cells leading to undetectable minimal residual disease. Thus the investigators expect to assess the safety and efficiency of pioglitazone in combination with imatinib mesylate in clinical trials. Maybe the combination therapy induce more patients in a detectable molecular response into a deeper molecular response. Furthermore, pioglitazone may be extensively adapted into the treatment of chronic phase chronic myelogenous leukemia patients as a common protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Treatment with imatinib mesylate for more than 2 years.
3. Patients with chronic phase chronic myelogenous leukemia having a complete cytogenetic response and a stable molecular response without complete molecular response.
4. Normal important organs such as kidney, liver and heart.

Exclusion Criteria:

1. Severe important organs disfunction such as liver and kidney.
2. Cardiovascular disease.
3. Osteoporosis in therapy.
4. Severe fluid retention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the rate of complete molecular response after the treatment of pioglitazone in combination with imatinib mesylate | one year

SECONDARY OUTCOMES:
the time for patients to complete molecular response from the beginning of adding pioglitazone | one year
the incidence rate of severe side effect or complication | one year

CONTACTS AND LOCATIONS:
Overall Officials: Li Meng, Study Chair — department of hematology, Wuhan Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prost S, Relouzat F, Spentchian M, Ouzegdouh Y, Saliba J, Massonnet G, Beressi JP, Verhoeyen E, Raggueneau V, Maneglier B, Castaigne S, Chomienne C, Chretien S, Rousselot P, Leboulch P. Erosion of the chronic myeloid leukaemia stem cell pool by PPARgamma agonists. Nature. 2015 Sep 17;525(7569):380-3. doi: 10.1038/nature15248. Epub 2015 Sep 2. PMID 26331539